CLINICAL TRIAL: NCT07118605
Title: Exploring the Potential of Minimally Invasive Sagittal Split Ramus Osteotomy to Transform Patient Outcomes: A Randomized, Double-Blind, Controlled Split Mouth Study
Brief Title: Minimally Invasive Sagittal Split Ramus Osteotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, İbrahim Mert Erkan, resident, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2024/110
Record Dates: First submitted 2025-07-29; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Orthognathic Surgical Procedures
Keywords: minimally invasive; sagittal split ramus osteotomy; orthognathic surgery; patient outcomes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally Invasive Sagittal Split Ramus Osteotomy (Experimental)
  Interventions: Procedure: Minimally Invasive Sagittal Split Ramus Osteotomy
- Conventional Sagittal Split Ramus Osteotomy (Active Comparator)
  Interventions: Procedure: Conventional Sagittal Split Ramus Osteotomy

INTERVENTIONS:
Procedure: Minimally Invasive Sagittal Split Ramus Osteotomy — This procedure involves a limited mucosal incision and tunnel dissection technique combined with low and short osteotomy and minimal soft tissue manipulation. The goal is to reduce surgical trauma, edema, blood loss, and operative time while maintaining clinical effectiveness.
  Arms: Minimally Invasive Sagittal Split Ramus Osteotomy
Procedure: Conventional Sagittal Split Ramus Osteotomy — This procedure follows the traditional wide exposure technique with full-thickness mucoperiosteal flap elevation. This method is widely accepted and serves as the control for comparison.
  Arms: Conventional Sagittal Split Ramus Osteotomy

SUMMARY:
This randomized, double-blind, controlled, split-mouth clinical trial investigates the effects of two different surgical approaches - the conventional technique and a minimally invasive technique - during bilateral sagittal split ramus osteotomy (SSRO) for mandibular deformity correction. The study will be conducted at the Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, Erciyes University.

Each patient will receive both surgical techniques, randomly assigned to either side of the mandible. All procedures will be performed under general anesthesia by the same surgeon. Intraoperative outcomes including bleeding volume and operative time will be recorded. Postoperative evaluations will be conducted on day 1, weeks 1, 2, and 4, and at 3 months to assess pain and swelling.

This study aims to determine whether the minimally invasive SSRO technique can improve surgical efficiency and reduce postoperative morbidity compared to the conventional approach, without compromising treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent sagittal split ramus osteotomy for mandibular dentofacial deformity
* Patients classified as ASA I or II
* Patients over 18 years of age

Exclusion Criteria:

* Patients with uncontrolled diabetes
* Patients with metabolic bone diseases (e.g., hyperparathyroidism, Paget's disease)
* Patients with syndromic conditions (e.g., Pierre Robin syndrome, Treacher Collins syndrome)
* Patients who had previously undergone mandibular surgery due to trauma, tumors, or cysts and had sequelae involving the lower jaw

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Operative Time | Intraoperative period (from skin incision to final suture placement)
  Operative time will be measured in minutes, separately for the right and left sides, from the initial skin incision to the final suture placement, using a chronometer.
Bleeding | Intraoperative period (from skin incision to final suture placement)
  Bleeding volume will be measured in milliliters from the initial skin incision to the final suture placement, using separate calibrated aspirators for the left and right sides.

SECONDARY OUTCOMES:
Postoperative Edema | Postoperative days 1, 7, 14, and 30
  The 3dMD imaging system (3dMD, Atlanta, GA) and 3dMD Vultus software were used to evaluate the amount of postoperative edema. Three-dimensional images were taken with the teeth in maximum intercuspation, lips relaxed, and eyes open on postoperative days 1, 7, 14, 30, and 90. Edema was calculated separately for the right and left sides and was recorded as surface area in square centimeters (cm²).
Postoperative Pain | Postoperative hours 1, 2, 4, 6, 8, 10, and 12
  Postoperative pain was evaluated using the Visual Analogue Scale for the right and left sides separately. In this scale, '0' meant no pain, and '100' represented maximum pain. Patients were questioned at postoperative 1st, 2nd, 4th, 6th, 8th, 10th, and 12th hours, and the results were recorded in the patient follow-up form.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Faculty of Dentistry Department of Oral and Maxillofacial Surgery, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No